CLINICAL TRIAL: NCT02181283
Title: Preventing Alcohol/Prescribed Drug Misuse in the National Guard: Web and Peer BI
Brief Title: MiSSION STRONG - Preventing AOS Misuse in the National Guard
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Frederic C. Blow, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AA023122; 1R01AA023122-01 (NIH)
Record Dates: First submitted 2014-06-26; First posted 2014-07-03 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: AOD Misuse
Keywords: alcohol; prescribed drugs; National Guard

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- W+W (Active Comparator): Web-delivered alcohol/prescribed drug misuse brief intervention with Web booster sessions (W+W).
  Interventions: Behavioral: W+W
- W+P (Active Comparator): Web-delivered brief intervention with Peer-delivered booster sessions (W+P).
  Interventions: Behavioral: W+P
- Enhanced Usual Care (No Intervention): Enhanced usual care.

INTERVENTIONS:
Behavioral: W+W — Web-delivered brief intervention: Participants receive a 30-40 minute Web-based intervention which includes a tailored review of participants' goals/values, feedback regarding their present alcohol/prescribed opioid/sedative use patterns and consequences, developing a discrepancy between their alcohol or prescribed drug use, ability to meet goals and values through a decisional balance exercise, and formulation of a tailored "change plan".
  Web booster sessions: Web boosters will be completed at 1, 2 and 3 months post-BI. Content is tailored to the individual based on answers to baseline questions and responses during Web-based BI. Web-based Booster will: 1) briefly ascertain current AOS use, 2) changes in AOS since completing Web BI, 3) progress toward goals, and 4) plans and encouragement for next steps.
  Other Names: Web-delivered brief intervention with Web booster sessions
  Arms: W+W
Behavioral: W+P — Web-delivered brief intervention: Participants receive a 30-40 minute Web-based intervention which includes a tailored review of participants' goals/values, feedback regarding their present alcohol/prescribed opioid/sedative use patterns and consequences, developing a discrepancy between their alcohol or prescribed drug use, ability to meet goals and values through a decisional balance exercise, and formulation of a tailored "change plan".
  Peer booster sessions: The peer supporter will work with participants at 1, 2, and 3 months post-Web-based BI. Peer supports will address Service Members' own goals and will provide emotional and informational support.
  Other Names: Web-delivered brief intervention with Peer-delivered booster sessions
  Arms: W+P

SUMMARY:
National Guard members, especially those who have been combat-deployed, are at high risk for developing alcohol- and prescription-related drug problems. The use of novel Web-based interventions combined with either Web-based boosters or Peer support sessions, may have a major public health impact for the National Guard by reducing hazardous use of alcohol of prescription drugs. The aims of the study are to develop, refine and test tailored motivational Brief Interventions (BIs) with varied continuing booster reinforcements (Web vs. Peer) and to conduct a randomized controlled trial comparing the efficacy of these BIs (W+W; W+P) to usual care on subsequent alcohol/drug consumption and consequences, including injury, mental and physical-health functioning, and HIV risk behaviors at 4-, 8-, and 12-months post-enrollment.

DETAILED DESCRIPTION:
The proposed study will test the efficacy of an easy-to-use, <40-minute, state-of-the-art tailored Web-based SBIRT (Screening, Brief Intervention, and Referral to Treatment) intervention combined with subsequent Web- or Peer-based boosters, compared to enhanced usual care (EUC). All participants will also receive a booklet with prevention information that includes general alcohol, opioid, and sedative use information as well as other health behaviors. The proposed study will screen ~ 4,300 unique Service Members as part of Soldier Readiness Processing in the Michigan National Guard (NG) to enroll 750 participants within 35 armories with alcohol and/or prescribed opioid or sedative misuse (AOS misuse). We will identify AOS misuse with a combination of the Alcohol Use Disorders Identification Test-Consumption (AUDIT-C) and an adapted version of the Pain Medication Questionnaire (PMQ). Computerized screening with touch-screen computer tablets will be used to recruit NG Service Members with AOS misuse in the prior 4 months. Participants will be randomized to one of three conditions:1) Web-delivered alcohol/prescribed drug misuse brief intervention with Web booster sessions (1/month for 3 months; W+W; n=250); 2) Web-delivered brief intervention with Peer-delivered booster sessions (at least 1/month for 3 months; W+P; n=250); or 3) Enhanced Usual Care (EUC; n=250). Random assignment will be stratified by gender and alcohol vs. prescription opioid/sedative misuse.

ELIGIBILITY:
Inclusion Criteria:

Individuals will be eligible to participate if they are in the Michigan Army National Guard and their unit is selected to participate in the proposed study. Individuals will be eligible to participate in the randomized trial if they:

* have an AUDIT-C score of 5 or more for men and 4 or more for women in the prior 4 months, indicating that they meet criteria for at-risk drinking/alcohol misuse; and/or
* use of prescribed opioids or sedatives in the prior 4 months in a manner that was inconsistent with their prescribed course of treatment (medical misuse: determined by items from an adapted PMQ).

Exclusion Criteria:

* under 18 years of age
* inability to speak and understand English
* inability to give informed, voluntary consent
* do not have access to the Web (e.g. home, work, library, WiFi-enabled tablet PCs (iPad), etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 757 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Alcohol use | change over time (4-, 8- and 12-months post baseline)
  The full AUDIT which includes the AUDIT-C, will be used to assess alcohol use. Quantity and frequency is measured by number of drinking days, number of drinks per day and number of binge drinking days. Alcohol related consequences are measured using the modified SIP.
Medical misuse of opioids or sedatives | change over time (4-, 8- and 12-months post baseline)
  Quantity and frequency is measured by number of days misused, and the NIDA-Modified ASSIST and adapted Pain Medication Questionnaire (PMQ) are used to assess medical misuse of prescribed opioids and medical misuse of prescribed sedatives. Consequences are measured using the modified SIP.

SECONDARY OUTCOMES:
Consequences of AOS use, including a) injury, b) mental and physical health functioning, and c) HIV-risk behaviors | 4-, 8- and 12-months post baseline
  3a) Injury is measured using the Revised Injury Behavior Checklist (RIBC). 3b) Mental and physical health functioning is measured using a brief version of the Short Form Health Survey (SF-12), the Generalized Anxiety Disorder (GAD-7) questionnaire, the Patient Health Questionnaire (PHQ), the Post-Traumatic Disorder Checklist-Military Version (PCL-5) and items from the Unit Risk Inventory, developed by the Army Substance Abuse Program.
  3c) HIV-risk behaviors are measured using questions from the HIV Risk-Taking Behavior Scale (HRBS).

CONTACTS AND LOCATIONS:
Overall Officials: Frederic C Blow, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blow FC, Walton M, Ilgen M, Ignacio RV, Walters H, Massey L, Barry KL, McCormick R, Coughlin LN. Peer- and web-based interventions for risky drinking among US National Guard members: Mission Strong randomized controlled trial. Addiction. 2023 Jul;118(7):1246-1257. doi: 10.1111/add.16172. Epub 2023 Apr 11. PMID 37041669
- [Derived] Coughlin LN, Blow FC, Walton M, Ignacio RV, Walters H, Massey L, Barry KL, McCormick R. Predictors of Booster Engagement Following a Web-Based Brief Intervention for Alcohol Misuse Among National Guard Members: Secondary Analysis of a Randomized Controlled Trial. JMIR Ment Health. 2021 Oct 26;8(10):e29397. doi: 10.2196/29397. PMID 34698652